CLINICAL TRIAL: NCT00722072
Title: A Phase II Open-Label Study of Sorafenib Plus Fulvestrant as Salvage Therapy for Hormone Receptor Positive Metastatic Breast Cancer Failing Prior Aromatase Inhibitor Treatment
Brief Title: Sorafenib and Fulvestrant in Treating Patients With Locally Advanced or Metastatic Breast Cancer That Did Not Respond to Aromatase Inhibitor Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor pulled funding and low accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004318; P30CA069533 (NIH); OHSU-4318; BAYER-OHSU-4318; CDR0000601002 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-07-24; First posted 2008-07-25 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Fulvestrant; Sorafenib

ARMS (1):
- Fulvestrant/ Sorafenib (Experimental): Fulvestrant: A loading dose will be administered intramuscularly to all subjects during cycle 1 of treatment as follows:
  * 500 mg IM on Day 1
  * 250 mg IM on Day 15 Upon completion of the loading dose, a fixed dose of Fulvestrant 250 mg IM will be administered on day 1 of the next 28 day cycle and every consecutive cycle until tumor progression or unacceptable toxicity occurs requiring discontinuation.
  Sorafenib: Subjects will take Sorafenib 800 mg/day administered as 400 mg bid (twice daily)each morning and evening approximately 12 hours apart. Treatment will begin on Day 1 of the study and continue daily until tumor progression or until unacceptable toxicity occurs.
  Interventions: Drug: fulvestrant; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: fulvestrant — Loading dose for cycle 1: 500 mg intramuscular(IM) on Day 1;250 mg IM on Day 15 Upon completion of the loading dose, a fixed dose of fulvestrant 250 mg IM will be administered on day 1 of the next 28 day cycle and every consecutive cycle until tumor progression or until unacceptable toxicity occurs requiring discontinuation of study therapy
Drug: sorafenib tosylate — Subjects will take sorafenib 800 mg/day administered as 400 mg bid (twice daily) each morning and evening approximately 12 hours apart. Treatment will begin on Day 1 of the study and continue daily until tumor progression or until an unacceptable toxicity occurs which would require delay, modification or discontinuation of study therapy

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving sorafenib together with fulvestrant may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sorafenib together with fulvestrant works in treating patients with locally advanced or metastatic breast cancer that did not respond to aromatase inhibitor therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the clinical activity of sorafenib tosylate and fulvestrant, as determined by a 4-month progression-free survival rate, in patients with hormone receptor-positive locally advanced or metastatic breast cancer that progressed after prior treatment with an aromatase inhibitor.

Secondary

* To determine the objective response rate in patients treated with this regimen.
* To determine the median time to progression in patients treated with this regimen.
* To determine the progression-free survival of patients treated with this regimen.
* To determine the overall survival of patients treated with this regimen.
* To establish the safety and tolerability profile of this regimen in these patients.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 1-28. Patients also receive fulvestrant intramuscularly on days 1 and 15 of course 1 and on day 1 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28-56 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of incurable breast cancer

  * Locally advanced or metastatic disease
* Measurable or evaluable disease

  * Measurable disease is defined as ≥ 1 uni-dimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral computed tomography(CT) scan

    * Bone-only metastases that can be imaged with bone scan AND magnetic resonance imaging (MRI) or bone scan AND plain x-ray is considered measurable disease
    * Tumor lesions that are situated in a previously irradiated area are considered measurable only if they are progressing at the time of study entry
  * Evaluable disease includes unresectable skin/chest wall metastases that can be photographed and whose size can be measured with a ruler

    * Bone-only metastases that can only be imaged using bone scan or malignant pleural effusion(s) only are not considered evaluable disease
* Previously treated with a third-generation aromatase inhibitor (e.g., letrozole, anastrazole, or exemestane) AND meets one of the following criteria:

  * Progressed during palliative aromatase inhibitor therapy
  * Recurred during adjuvant aromatase inhibitor therapy
  * Recurred within 12 months of completing adjuvant aromatase inhibitor therapy
* Human Epidermal growth factor Receptor 2(HER2/neu)-negative tumor

  * No Human Epidermal growth factor Receptor 2(HER2/neu) overexpression (i.e., tumor staining 3+ by immunohistochemistry [IHC] or gene amplified by Fluorescence In Situ Hybridization [FISH])
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive, defined as ≥ 10% of malignant cells with positive nuclear staining

PATIENT CHARACTERISTICS:

* Postmenopausal
* Eastern Cooperative Group(ECOG) performance status 0-1
* Life expectancy ≥ 16 weeks
* Neutrophil count ≥ 1,500/mm^³
* Platelet count ≥ 100,000/mm^³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine < 2 mg/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase(AST) ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* International Normalized Ratio(INR) < 1.5 OR Prothrombin time/ partial thromboplastin time (PT/PTT) normal
* Left ventricular ejection fraction(LVEF) normal by Multiple Gated Acquisition(MUGA) or ECHO
* No known allergy to sorafenib tosylate or fulvestrant
* No cardiac disease, including any of the following:

  * New York Heart Association(NYHA) class III-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest) or new-onset angina (within the past 3 months)
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg despite optimal medical management
* No thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attacks), within the past 6 months
* No known HIV infection or chronic hepatitis B or C infection
* No infection that requires IV antibiotics or produces a fever > 100°F within the past 72 hours
* No pulmonary hemorrhage/bleeding event ≥ Common terminology criteria for adverse events(CTCAE) grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 2 weeks
* No serious, nonhealing wound, ulcer, or bone fracture
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption problem
* No second malignancy within the past 5 years, except adequately treated and cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No underlying medical condition that, in the principal investigator's opinion, will make the administration of study drug hazardous or would obscure the interpretation of adverse events

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for metastatic or unresectable locally advanced breast cancer
* No prior sorafenib tosylate or other Vascular endothelial growth factor(VEGF)-targeting therapies
* More than 2 weeks since prior major surgery or open biopsy
* No concurrent anticoagulation with warfarin or heparin
* No concurrent Hypericum perforatum (St. John wort) or rifampin
* No other concurrent anticancer agents, including chemotherapy or biological therapy
* No other concurrent investigational drugs
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chui, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib and Fulvestrant: Fulvestrant:Will be administered to the subject intramuscularly. Administered to all subjects during cycle 1 of treatment as follows:
  * 500 mg IM on Day 1
  * 250 mg IM on Day 15
  Sorafenib: 800 mg/day administered as 400 mg bid (twice daily) each morning and evening approximately 12 hours apart. Treatment will begin on Day 1 of the study and continue daily until tumor progression or until an unacceptable toxicity occurs which would require delay, modification or discontinuation of study therapy.
Period: Overall Study
Arm/Group | Sorafenib and Fulvestrant
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.166 (9.0235)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival at 4 Months
Description: Progression-free survival rate is defined as the proportion of subjects who are progression free (CR, PR and SD) at 4 months after initiating treatment with sorafenib plus fulvestrant. Complete Response (CR):Disappearance of all target (both measurable and evaluable)lesions. Partial Response (PR):At least a 30% decrease in the sum of the longest diameter (LD) of both measurable and evaluable target lesions. Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease(PD).
Time Frame: 4 months after initiating treatment with sorafenib plus fulvestrant.
Measure: Number; unit: Participants
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 12
Participants | 6

2. Secondary Outcome: Objective Response Rate
Time Frame: Every 8 weeks (two cycles) while receiving study therapy.
Population: Response assessment data was not collected past 4 months due to early study termination.
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression
Time Frame: Start of treatment to time of progression.
Population: Progression data was not collected due to early study termination.
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: Start of treatment to time of progression or death, whichever comes first.
Population: Long term survival data was not collected due to early study termination
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: 28 to 56 days after discontinuation of study therapy
Population: Long term survival data was not collected due to early study termination
Arm/Group | Sorafenib and Fulvestrant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib and Fulvestrant
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib and Fulvestrant (N=9)
Hand-foot syndrome (HFS) (General disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Desquamation (Skin and subcutaneous tissue disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib and Fulvestrant (N=9)
Neutropenia (Blood and lymphatic system disorders) | 9
Myalgias (Musculoskeletal and connective tissue disorders) | 9
Arthralgias (Infections and infestations) | 9
Fatigue (General disorders) | 9
Pruritis (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No